CLINICAL TRIAL: NCT06571214
Title: An Exploratory, Randomized, Open-label, Controlled Study to Evaluate the Potential Benefit of r-hLH Addition in Patients Aged 35 to 40 Under Ovarian Stimulation Treatment
Brief Title: Potential Benefit of r-hLH Addition in Patients Aged 35 to 40 Under Ovarian Stimulation Treatment
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Nanjing University (Other)
Responsible Party: Principal Investigator, Li-jun Ding, Director of Reproductive Medicine Department, Nanjing University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MS700642_0020
Record Dates: First submitted 2024-08-05; First posted 2024-08-26 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Infertility
Keywords: recombinant human LH; recombinant human FSH; ovarian stimulation treatment; advanced maternal age population
MeSH Terms: conditions — Infertility | interventions — Injections; follitropin alfa; Luteinizing Hormone, beta Subunit

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): The r-hFSH starting dose will be based on the patient's profile and physician's experience. r-hLH will be added at a ratio of 2:1 starting from day 1 of r-hFSH administration; the dose of r-hFSH during COS will be adjusted by the physician based on clinical experience and the patient's ovarian response, and the r-hFSH: r-hLH dose will be 2:1, continuing to 24~48 hours prior to trigger drug injection.
  For both groups, daily injection of 0.25 mg of cetrorelix (Cetrotide®, Merck Serono S.A.) will be administrated subcutaneously when at least one follicle with diameter ≥ 14 mm or serum LH level exceeds 10 IU/L or LH level is 2 folder than basal LH level or P level exceeds 0.8 ng/ml, continuing until ovulation triggering day. Cetrorelix can be administrated earlier in patients with advanced age or diminished ovarian reserve according to judgment of clinicians.
  Interventions: Drug: Recombinant Human Follitropin Alfa Solution for Injection (Gonal-f®); Drug: Recombinant Human Lutropin alfa for Injection (r-hLH, Luveris®)
- Control group (Active Comparator): r-hFSH alone will be administrated for ovarian stimulation. The r-hFSH starting dose will be based on the patient's profile and physician's experience. The dose of r-hFSH during COS will be adjusted by the physician based on clinical experience and the patient's ovarian response, continuing to 24~48 hours prior to trigger drug injection.
  For both groups, daily injection of 0.25 mg of cetrorelix (Cetrotide®, Merck Serono S.A.) will be administrated subcutaneously when at least one follicle with diameter ≥ 14 mm or serum LH level exceeds 10 IU/L or LH level is 2 folder than basal LH level or P level exceeds 0.8 ng/ml, continuing until ovulation triggering day. Cetrorelix can be administrated earlier in patients with advanced age or diminished ovarian reserve according to judgment of clinicians.
  Interventions: Drug: Recombinant Human Lutropin alfa for Injection (r-hLH, Luveris®)

INTERVENTIONS:
Drug: Recombinant Human Follitropin Alfa Solution for Injection (Gonal-f®) — As a r-hFSH agent, Gonal-f® is used for COS. It is a prefilled ready to use pen device containing follitropin alfa for injection and is designed for subcutaneous self-administration by patients undergoing COS for ART. It is available as dose presentations of 150 IU and 450 IU. The investigators and/or his/her delegate/s will explain the use of Gonal-f® prefilled pen. Gonal-f® will be prescribed by the investigator based on clinical diagnosis and treatment routines, and will not be provided free of charge.
  Arms: Treatment group
Drug: Recombinant Human Lutropin alfa for Injection (r-hLH, Luveris®) — This product is a white freeze-dried powder and a colorless and clear injection solvent, and stored away from light under 25℃ in the original packaging. Luveris® will be provided free of charge.

SUMMARY:
This will be an exploratory, prospective, randomized, open-label and controlled trial to evaluate the potential benefit of r-hFSH:r-hLH 2:1 co-treatment starting from COS D1 versus r-hFSH alone in patients aged 35 to 40 under ovarian stimulation treatment.

After signing informed consent form (ICF), all eligible participants will be randomly assigned in a 1:1 ratio to either treatment or control group, and GnRH antagonist protocol will be used in both treatment and control groups.

DETAILED DESCRIPTION:
This will be an exploratory, prospective, randomized, open-label and controlled trial to evaluate the potential benefit of r-hFSH:r-hLH 2:1 co-treatment starting from COS D1 versus r-hFSH alone in patients aged 35 to 40 under ovarian stimulation treatment.

After signing informed consent form (ICF), all eligible participants will be randomly assigned in a 1:1 ratio to either treatment or control group, and GnRH antagonist protocol will be used in both treatment and control groups.

1. Treatment group: The r-hFSH starting dose will be based on the patient's profile and physician's experience. r-hLH will be added at a ratio of 2:1 starting from day 1 of r-hFSH administration; the dose of r-hFSH during COS will be adjusted by the physician based on clinical experience and the patient's ovarian response, and the r-hFSH: r-hLH dose will be 2:1, continuing to 24~48 hours prior to trigger drug injection.
2. Control group: r-hFSH alone will be administrated for ovarian stimulation. The r-hFSH starting dose will be based on the patient's profile and physician's experience. The dose of r-hFSH during COS will be adjusted by the physician based on clinical experience and the patient's ovarian response, continuing to 24~48 hours prior to trigger drug injection.

The estimated treatment duration is 11 days from the first day of COS until 24~48 h prior to trigger drug injection, and this may vary depending on individual circumstances.

Follicular development, serum E2 and P levels will be monitored during COS according to the investigator site's ART practice until the criteria to administer trigger drug are met to induce final oocyte maturation. Trigger drug administration is to be performed according to the site's routine clinical practice.

Oocyte pick-up (OPU), IVF/ICSI, ET, and luteal phase support (LPS) will be performed according to the site's routine practice. LPS will be started after oocyte retrieval in fresh embryo transfer.

ELIGIBILITY:
Inclusion Criteria:

* Age 35 to 40 (including 40)
* 18.5<BMI<28 kg/m2
* AFC up to 14
* First or second ART cycle
* Planned for ovarian stimulation with GnRH-antagonist for down-regulation
* Ejaculated sperm

Exclusion Criteria:

* Contraindications to ART treatment
* History of two or more spontaneous miscarriages
* History of two or more implantation failures after fresh or frozen-warmed embryo transfers
* Diagnosis of severe endometriosis
* Patients with endocrine and metabolic diseases (diabetes mellitus, hypogonadotropic amenorrhea, genital system tumors, hyperprolactinemia, etc.)
* Confirmed chromosomal abnormalities

Ages: 35 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Patients aged 35 to 40 under ovarian stimulation treatment
Enrollment: 300 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Good quality embryo rate (cleavage stage) | Day 3 after fertilization
  Cleavage stage good-quality embryos are defined as embryos derived from normally fertilized zygotes with 7~9 cells on day 3 post-fertilization, stage-specific cell size, less than 10% fragmentation, and no multinucleation. Cleavage stage good-quality embryo rate is defined as the number of cleavage stage good-quality embryos divided by the number of normally fertilized zygotes. Embryos will be assessed by two independent experienced embryologists to minimize intra-observation variability.

SECONDARY OUTCOMES:
Number of oocytes | 24 hours after Oocytes pick up
  Number of oocytes is defined as the total number of oocytes obtained through transvaginal ultrasound guided puncture on the day of OPU. All follicles with an estimated diameter of ≥12 mm should be punctured.
Number of MII oocytes (analyzed in ICSI subgroup only) | 24 hours after Oocytes pick up
  Number of MII oocyte is defined as the total number of an oocyte at metaphase of meiosis II, exhibiting the first polar body and with the ability to become fertilized
Total r-hFSH dose | 24 hours after ovulation triggering
  Total r-hFSH dose is defined as the total dose of r-hFSH used for subcutaneous injection during COS period.
Fertilization rate | 24 hours after fertilization
  * IVF normal fertilization rate is defined as the number of oocytes with 2PN and 2PB divided by the number of COCs inseminated.
  * ICSI normal fertilization rate is defined as the number of oocytes with 2PN and 2PB divided by the number of MII oocytes injected.
Blastocyst development rate | 5 days after fertilization, up to 7 days
  Blastocyst development rate is defined as the proportion of blastocysts observed at 116 ± 2 h post-insemination as a function of the number of normally fertilized oocytes.
Utilizable embryo rate | 5 days after fertilization, up to 7 days
  Utilizable embryo rate is defined as the number of embryos (or blastocysts) suitable for transfer or cryopreservation as a function of the number of normally fertilized (2PN) oocytes observed on Day 1.
Implantation rate | At 4-6 weeks of amenorrhea after customized timing of embryo transfer
  Implantation rate is defined as the number of gestational sacs observed divided by the number of embryos transferred using transvaginal ultrasound 4~6 weeks after embryo transfer.
Clinical pregnancy rate (per transfer cycle and per oocyte retrieval cycle) | At 4-6 weeks of amenorrhea after customized timing of embryo transfer
  Clinical pregnancy rate is defined as the number of clinical pregnancies expressed per 100 initiated cycles, aspiration cycles, or embryo transfer cycles. Clinical pregnancy is defined as the presence of gestational sac (intrauterine or ectopic) using ultrasound examination at 4~6 weeks after embryo transfer.
Ongoing pregnancy rate | At 12 weeks of amenorrhea after customized timing of embryo transfer
  Ongoing pregnancy rate is defined as the number of intrauterine pregnancies continued for 12 gestational weeks divided by the number of embryo transfer cycles.
Ovarian sensitivity index (OSI) | 24 hours after fertilization
  OSI is defined as the total r-hFSH dose divided by the number of oocytes retrieved.
Follicular output rate (FORT) | 24 hours after fertilization
  FORT is defined as the number of pre-ovulatory follicles (16~22 mm) on the day of trigger divided by the AFC (3~8 mm)
Follicle oocyte index (FOI) | 24 hours after fertilization
  FOI is defined as the number of total oocytes retrieved divided by the AFC
Safety Assessments | During the COS cycle (average cycle range 11 days), Up to 12 weeks after transfer
  AE, SAE and OHSS

CONTACTS AND LOCATIONS:
Overall Officials: Haiming Xia, Dr., Principal Investigator — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (1):
- Nanjing Drum Tower Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No